CLINICAL TRIAL: NCT00380289
Title: Early Metabolic Changes With Thiazide or Beta Blocker Therapy for Essential Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OGTT1
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2006-09-25 (Estimated); Status verified 2006-09

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; Glucose metabolism; Thiazides; Beta blockers
MeSH Terms: conditions — Essential Hypertension | interventions — Thiazides; Adrenergic beta-Antagonists

INTERVENTIONS:
Drug: Thiazide and beta blocker

SUMMARY:
Can the oral glucose tolerance test detect changes after 4 weeks treatment with thiazide diuretics or beta blockers or combination of the two?

DETAILED DESCRIPTION:
We will be comparing the two most commonly used drugs to treat hypertension, atenolol and bendrofluazide, in patients for whom the drugs (and the doses to be used) are licenced.

We propose an initial open label pilot study of 10-12 patients to confirm final doses to be tested, the duration of therapy for optimum timing of the OGTT and tolerability of doses selected. The pilot study will also be used to confirm sample size calculations for the main study.The protocol for the pilot study will be identical to the main study, but there will not be a placebo phase and the treatment will not be blinded.

The main study will be double-blind, placebo controlled, cross-over study, of approximately 66 patients in which each patient receives in random order, 4 weeks treatment with either Bendrofluazide 5-10mg daily, Atenolol 50-100mg daily or combination of Bendrofluazide 2.5-5mg and Atenolol 25-50mg daily. There will be a forced titration from the lower to the higher dose stated half way through each dosing period. There will be a 1 month placebo wash-out between each dosing period.

At 0, 2 and 4 weeks of each treatment phase, patients will attend the Clinical Investigation Ward (CIW), fasting, for performance of an oral glucose tolerance test (OGTT). Blood will be drawn from an intravenous cannula, for the measurements of glucose and insulin at 0, 0.5, 1 and 2 hours.

Blood pressure will be measured at each study visit using an Omron machine. The patients will also be given a blood pressure machine to take home and will be asked to measure and record their blood pressure at least twice per week. If their blood pressure is under 110/70mmhg or over 160/110mmHg at any time or if the patient has symptoms e.g. headache or dizziness, the patient will be asked to contact study staff. If the blood pressure remains over 160/110 for two measurements, then another antihypertensive therapy may be commenced, or the patient withdrawn from the study. If blood pressure is < 110/70 mmHg with symptoms then a decision may be made to terminate their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers will be aged 18-75 years.
* Hypertension- either

  * untreated, BP 140-170/90-110
  * treated for over 1 month with drugs other than beta blockers or diuretic and BP>140/85
  * treated for over 1 month with drugs other than beta blockers or diuretic and BP<140/85 and patient willing to change medication for eight months.

Exclusion criteria:

* Any patient already taking thiazide diuretics or beta blockers in whom these drugs cannot be switched to alternative drugs with similar or better blood pressure control.
* Any patient who is intolerant of these medications will be excluded from the study.
* Patients with gout, asthma or any other contraindications to the study drugs will be excluded.
* Women of child bearing age not using contraception.
* Volunteers with heart failure, liver failure, renal failure, terminal illnesses (e.g. cancer)
* Volunteers not able to give informed consent
* Patients with diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2006-09

PRIMARY OUTCOMES:
Can the oral glucose tolerance test detect changes after 4 weeks treatment with thiazide diuretics or beta blockers or combination of the two?

SECONDARY OUTCOMES:
Do patients show a similar change in glucose tolerance after thiazide or beta blocker therapy?
Does the combination of drugs cause a greater reduction in glucose tolerance than expected from the response to each drug taken alone?

CONTACTS AND LOCATIONS:
Overall Officials: Professor MJ Brown, MA MSC MD FRCP, Principal Investigator — Addenbrookes Hosptal NHS Trust/ University of Cambridge
Locations (1):
- Clinical Pharmacology Unit, Box 110, Level 3 ACCI, Addenbrookes Hospital, Cambridge, United Kingdom

REFERENCES:
- [Derived] Stears AJ, Woods SH, Watts MM, Burton TJ, Graggaber J, Mir FA, Brown MJ. A double-blind, placebo-controlled, crossover trial comparing the effects of amiloride and hydrochlorothiazide on glucose tolerance in patients with essential hypertension. Hypertension. 2012 May;59(5):934-42. doi: 10.1161/HYPERTENSIONAHA.111.189381. Epub 2012 Apr 9. PMID 22493073